CLINICAL TRIAL: NCT05720533
Title: Safety and Efficacy of Disitamab Vedotin Combined With Sintilimab as First-line Treatment of Elderly Patients With HER2 Overexpression Gastric Cancer
Brief Title: Disitamab Vedotin Combined With Sintilimab as First-line Treatment of Elderly Patients With Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20221383
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin Combined With Sintilimab (Experimental): Treatment regimen is Disitamab vedotin 2.5mg/kg and Sintilimab 200mg every 21 days, until disease progression or intolerable adverse reactions or death.
  Interventions: Drug: Disitamab Vedotin Combined With Sintilimab

INTERVENTIONS:
Drug: Disitamab Vedotin Combined With Sintilimab — Disitamab Vedotin injection：2.5mg/kg，IV，Q3W Sintilimab injection：200mg，IV, Q3W
  Other Names: Combined treatment group

SUMMARY:
This study aims to explore the safety and efficacy of Disitamab vedotin combined with Sintilimab in elderly patients with HER2 overexpression Gastric Cancer. This is a single-arm exploratory clinical study. 20 patients with eHER2 overexpression gastric cancer are scheduled to be enrolled. Treatment regimen is Disitamab vedotin 2.5mg/kg and Sintilimab 200mg every 21 days, until disease progression or intolerable adverse reactions or death.

DETAILED DESCRIPTION:
The primary objective of this study was to explore the safety and median PFS of Disitamab vedotin combined with Sintilimab as first-line treatment in elderly patients with HER2 overexpression Gastric Cancer.The secondary objective of this study was to evaluate the ORR, DCR, DOR and OS of Disitamab vedotin combined with Sintilimab as first-line treatment in elderly patients with HER2 overexpression Gastric Cancer.To provide a better treatment plan for elderly patients with Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) Volunteer to take part in the study ;
* 2) Age ≥65 , male or female;
* 3) Gastric cancer or adenocarcinoma of gastroesophageal junction confirmed by histology and/or cytology;
* 4) Have not received systematic treatment; If the subject has received adjuvant therapy after completing radical treatment for early gastric cancer and the subject has relapsed disease, ensure that the end of adjuvant therapy is more than 6 months from the first dose of the study and that various toxicities due to the adjuvant therapy have recovered.
* 5) The HER2 immunohistochemistry (IHC) test result is IHC 3+or 2+, and the previous test results of the subject (confirmed by the investigator) are acceptable;
* 6) At least one assessable lesion (RECIST 1.1 );
* 7) Expected survival time ≥ 6 months;
* 8) ECOG 0-2;
* 9) If the main organs function normally, they meet the following standards:

Blood routine examination (no blood transfusion and G-CSF use within 14 days before screening):

1. Hemoglobin ≥ 90 g/L;
2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L；
3. White blood cell count ≥ 3.0 × 109/L；
4. Platelet count ≥ 80 × 109/L；

   Blood biochemical examination (albumin was not used within 14 days before screening):
5. Albumin ≥ 28 g/L;
6. Total bilirubin ≤ 2 × Upper limit of normal value (ULN);
7. In the absence of liver metastasis, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 2.5 × ULN； ALT, AST and ALP ≤ 5× ULN in case of liver metastasis ；
8. Alkaline phosphatase (ALP) ≤ 5 × ULN；
9. Creatinine ≤ 1.5 × ULN； Or the creatinine clearance rate (CrCl) calculated by Cockcroft Gault formula is ≥ 50 mL/min;

   Coagulation function:
10. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN；

j) Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN。

Exclusion Criteria:

* 1) Have a history of malignant tumors other than gastric cancer, except for the following two cases:

  1. The patient has received possible curative treatment and there is no evidence of the disease within 5 years;
  2. The resected skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ and other carcinoma in situ were successfully received;
* 2) Have received allogeneic stem cells or solid organ transplantation in the past;
* 3) Patients who have received other anti-tumor systemic therapy in the past (including traditional Chinese medicine with anti-tumor indications), and have been less than 4 weeks from the completion of treatment to the administration of this study, or the adverse events caused by previous treatment have not recovered to ≤ CTCAE level 1 (except hair loss and pigmentation);
* 4) Previous or current congenital or acquired immunodeficiency disease;
* 5) Allergic to the study drug;
* 6) Other significant clinical and laboratory abnormalities, which the researchers think affect the safety evaluation;
* 7) Serious infection in active period or poorly controlled clinically;
* 8) Not recovered from the operation;
* 9) Pregnant or lactating women, and women or men with fertility who are unwilling or unable to take effective contraceptive measures;
* 10) Other situations that the investigator thinks are not suitable for inclusion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free-Survival) | 24 months
  The time from randomization to tumor progression or death.The efficacy of this study was determined according to Recist version 1.1 criteria.

SECONDARY OUTCOMES:
ORR（Objective Response Rate） | 24 months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
DCR（Disease control rate） | 24 months
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
DOR（Duration of response） | 24 months
  DoR was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The time of the initial response was defined as the latest of the dates contributing toward the first visit response of CR or PR. If a patient did not progress following a response, then their DoR was censored at the PFS censoring time.
OS (Overall survival time) | 24 months
  The time of death from all causes for all patients from the date of randomization.
The Adverse Events | 24 months
  AEs are any adverse medical events that occur in a subject or clinical subject and is not necessarily causally related to the treatment. Safety assessment in this study was conducted by the investigator in accordance with the definition of CTCAE 5.0.

IPD SHARING:
Plan to Share IPD: No